CLINICAL TRIAL: NCT01047566
Title: The Effect of the Addition of Dronedarone to, Versus Increase of, Existing Conventional Rate Control Medication on Ventricular Rate During Persistent Atrial Fibrillation
Brief Title: Effect of Addition of Dronedarone to Standard Rate Control Therapy on Ventricular Rate During Persistent Atrial Fibrillation (AFRODITE)
Acronym: AFRODITE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DRONE_L_05066; 2009-018215-53 (EudraCT Number); NCT01117207 (obsolete NCT alias)
Record Dates: First submitted 2010-01-12; First posted 2010-01-13 (Estimated); Last update posted 2011-11-10 (Estimated); Status verified 2011-11

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Dronedarone; Adrenergic beta-Antagonists; Calcium Channel Blockers; Digoxin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Addition of dronedarone (Experimental): Addition of Dronedarone to existing rate control medication (beta blocker and/or calcium antagonist)
  Interventions: Drug: Dronedarone
- Dose Increase (Active Comparator): Dose increase of existing rate control medication (beta blocker or calcium antagonist or digoxin)
  Interventions: Drug: Beta blocker or calcium antagonist or digoxin

INTERVENTIONS:
Drug: Dronedarone — Pharmaceutical form: tablet Route of administration: oral Dose regimen: 400 mg twice daily for 12 weeks (+/- 5 days)
  Other Names: Multaq
  Arms: Addition of dronedarone
Drug: Beta blocker or calcium antagonist or digoxin — Dose increase of beta blocker or calcium antagonist or digoxin
  Arms: Dose Increase

SUMMARY:
The primary objective of this study is to:

Assess whether the addition of dronedarone to existing conventional rate control therapy leads to a reduced ventricular rate after 1 week in patients with a high Heart Rate (HR) at rest during Atrial Fibrillation (AF) in comparison to an increase of conventional therapy.

The secondary objectives of this study are to compare both study arms with regard to:

* Ventricular rate after 3 months
* Number of registered AF episodes
* Number of symptomatic AF episodes
* Severity of AF and AF-like symptoms
* Rate of premature study discontinuation
* Number of symptomatic episodes of bradycardia
* Incidence of low heart rate (<60 bpm)

ELIGIBILITY:
Inclusion Criteria:

* Persistent AF with HR >80 bpm at rest despite treatment with ≤ 2 rate control agents (i.e. beta blocker and/or calcium antagonist - Patients using digoxin are eligible)
* Documented AF in the past 24 hours
* Treated with the following rate control medication:
* beta blocker or
* calcium antagonist or
* beta blocker plus calcium antagonist or
* beta blocker plus digoxin or
* calcium antagonist plus digoxin
* Anticoagulant treatment in line with local guidelines

Exclusion Criteria:

* Incapacitated patients
* Paroxysmal or permanent AF
* Use of class I or III anti-arrhythmic drugs in the past 12 weeks
* Scheduled cardioversion or pulmonary vein ablation
* Unstable New York Heart Association (NYHA) class III and all class IV Heart Failure
* AV block grade 2 or 3
* Known severe renal impairment (serum creatinine > 180 μmol/l)
* Known severe hepatic impairment (AST, ALT > 3 x Upper Limit of Normal (ULN))
* Contra-indication for dronedarone
* Participation in a clinical drug study in the 3 months prior to inclusion
* Women of childbearing potential, who do not use adequate contraception
* Lactating women

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 46 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2010-04; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Ventricular rate | One week

SECONDARY OUTCOMES:
Ventricular rate | 12 weeks
Patients with registered AF episodes | Within the 12 weeks after randomization
Patients with symptomatic AF episodes | Within the 12 weeks after randomization
Severity of AF and AF-like symptoms | Within the 12 weeks after randomization
Premature study discontinuation | Within the 12 weeks after randomization
  Premature study discontinuation for all reasons including those where the patients must go off study prematurely as per protocol (ie. in case of cardioversion during the 1st study week, 2nd cardioversion after the 1st study week, addition of anti-arrhythmic drug, ablation or other surgical AF related intervention)
Patients with symptomatic episodes of bradycardia | Within the 12 weeks after randomization
Patients with low heart rate (<60 bpm) | Within the 12 weeks after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, PE Gouda, Netherlands